CLINICAL TRIAL: NCT01275586
Title: Pilot Study of Tasigna®/Nilotinib (AMN107) in Neurofibromatosis (NF1) Patients With Plexiform Neurofibromas
Brief Title: Study of Tasigna®/Nilotinib (AMN107) in Neurofibromatosis (NF1) Patients With Plexiform Neurofibromas
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-06; CAMN107YUS29T (Other: Novartis)
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Neurofibromatosis; NF1; Neurofibromas
Keywords: NF1; plexiform neurofibromas; nilotinib; Tasigna
MeSH Terms: conditions — Neurofibromatoses; Neurofibroma; Neurofibroma, Plexiform | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tasigna (Experimental): Following enrollment each subject will initially receive the drug Tasigna orally at 200 mg twice daily for two weeks. If tolerated, the dose will be increased to 300 mg twice daily after a minimum of two weeks and will be increase to a maximum dose of 400mg twice daily after an additional two weeks if tolerated. Subjects will have his/her dose increased as tolerated dose during the first three months of therapy. The maximum targeted dose is 400mg twice daily.
  Interventions: Drug: Tasigna

INTERVENTIONS:
Drug: Tasigna — Following enrollment each subject will initially receive Tasigna orally at 200 mg twice daily for two weeks. If tolerated, the dose will be increased to 300 mg twice daily after a minimum of two weeks and will be increase to a maximum dose of 400mg twice daily after an additional two weeks if tolerated.
  Other Names: Nilotinib

SUMMARY:
The purpose of this Pilot Study is to determine if NF1 patients with plexiform neurofibromas treated with Tasgina® respond to therapy.

DETAILED DESCRIPTION:
This is an open-label Pilot Study to determine the efficacy of Tasigna® in adults with neurofibromatosis (NF1) and plexiform neurofibromas with the secondary goals of determining the toxicity, and tumor markers in this genetically defined population. The rationale for this study arises from the response of human and murine NF1 cells to Tasigna® in vitro and the clinical response in NF1 patients with plexiform neurofibromas using the similar drug, Gleevec®. Following enrollment each subject will initially receive Tasigna orally at 200 mg twice daily for two weeks. If tolerated, the dose will be increased to 300 mg twice daily after a minimum of two weeks and will be increase to a maximum dose of 400mg twice daily after an additional two weeks if tolerated. Subjects will have his/her dose increased as tolerated dose during the first three months of therapy. The maximum targeted dose is 400mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > or = 18 years of age.
2. Clinical diagnosis of neurofibromatosis type 1 (NF1)
3. Presence of clinically significant plexiform neurofibromas (tumors that are potentially life threatening or are impinging on vital structures or significant impairment in the quality of life from pain or other symptoms)
4. Patients must have measurable disease by magnetic resonance imaging (MRI)(as defined by Response Evaluation Criteria in Solid Tumors, see Appendix 4)
5. Patients must have a Karnofsky Performance Status of ≥50%
6. Adequate end organ function, defined as the following:

   * Creatinine < 1.5 x ULN
   * ANC > 1.5 x 109/L
   * Platelets > 100 x 109/L
   * Total bilirubin < 1.5 x ULN

     - Does not apply to patients with isolated hyperbilirubinemia (e.g., Gilbert's disease) grade <3.
   * AST (SGOT) and ALT (SGPT) < 2.5 x ULN
   * Serum amylase and lipase ≤ 1.5 x ULN
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Patients must have the following laboratory values (WNL = within normal limits at the local institution lab) or corrected to within normal limits with supplements prior to the first dose of study medication:
   * Potassium (WNL)
   * Magnesium (WNL)
   * Phosphorus (WNL)
   * Calcium (WNL)

Exclusion Criteria:

1. Previous treatment with any other tyrosine kinase inhibitor
2. Impaired cardiac function including any one of the following:

   i. Inability to monitor the QT interval on ECG ii. Congenital long QT syndrome or a known family history of long QT syndrome. iii. Clinically significant resting brachycardia (<50 beats per minute) iv. QTc > 450 msec on baseline ECG. If QTc >450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc v. Myocardial infarction within 12 months prior to starting study vi. Other clinically significant uncontrolled heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension) vii. History or presence of clinically significant ventricular or atrial tachyarrhythmias
3. Patients currently receiving treatment with strong CYP3A4 inhibitors and treatment cannot be either discontinued or switched to a different medication prior to starting study drug. (Appendix 1).
4. Patients currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug (Appendix 3)
5. Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection or gastric bypass surgery).
6. Acute or chronic pancreatic disease
7. Patient has known brain metastasis. Non specific CNS changes on MRI characteristic with NF1 are allowed.
8. Another primary malignant disease, which requires systemic treatment (chemotherapy or radiation)
9. Acute or chronic liver disease or severe renal disease considered unrelated to the cancer.
10. History of significant congenital or acquired bleeding disorder unrelated to cancer
11. Major surgery within 4 weeks prior to Day 1 of the study or who have not recovered from prior surgery.
12. Treatment with other investigational agents within 30 days of Day 1.
13. History of non-compliance to medical regimens or inability to grant consent.
14. Female patients who are pregnant, breast feeding, or of childbearing potential without a negative pregnancy test prior to baseline. Male or female patients of childbearing potential unwilling to use contraceptive precautions throughout the trial and 3 months following discontinuation of study drug. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Women of childbearing potential must have a negative serum pregnancy test prior to the first dose of nilotinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Markel, MD, Study Chair — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tasigna
Started | 6
Completed | 3
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Tasigna
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Disease Response
Description: To estimate the disease control rate (PD,SD, PR, CR) with Tasigna® in patients with neurofibromas (NF1) using standard RECIST criteria. Complete Response (CR) is defined as; disappearance of all target lesions. Partial Response (PR) is defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as a reference the baseline sum longest diameter. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started. Disease Progression (PD) is defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tasigna
Number analyzed (Participants) | 3
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Stable Disease (SD) | 2
  Progressive Disease (PD) | 1

ADVERSE EVENTS:
Time Frame: adverse event data was collected while participants were on study treatment and for 30 days after last day of study treatment
Arm/Group | Tasigna
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasigna (N=6)
Elevated Lipase (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasigna (N=6)
Conjunctivitis (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
dyspepsia (Gastrointestinal disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
pain (General disorders) | 1 (1)
scrotal infection (Infections and infestations) | 1 (1)
Blood Bilirubin increased (Investigations) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 2 (2)
Elevated Amylase (Investigations) | 1 (1)
Elevated Lipase (Investigations) | 1 (1)
Weight Loss (Investigations) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Myalagia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in chest wall (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Join Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Bladder Infection (Renal and urinary disorders) | 1 (1)
Kidney Infection (Renal and urinary disorders) | 1 (1)
Bladder Spasm (Renal and urinary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes